CLINICAL TRIAL: NCT02520843
Title: An Innovative Treatment for Fistula-in-ano in Crohn Disease : Local Micro Reinjection of Autologous Fat and Stromal Vascular Fraction
Brief Title: An Innovative Treatment for Fistula-in-ano in Crohn Disease : Local Micro Reinjection of Autologous Fat and SVF
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-002602-31
Record Dates: First submitted 2015-08-05; First posted 2015-08-13 (Estimated); Last update posted 2019-01-17 (Actual); Status verified 2019-01

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Crohn's disease treated by SVF (Experimental): Patients with Crohn's disease and fistula-in-ano refractory to conventional medical and surgical treatment, treated by Stromal Vascular Fraction ( SVF) reinjection
  Interventions: Drug: stromal vascular fraction (SVF)

INTERVENTIONS:
Drug: stromal vascular fraction (SVF) — stromal vascular fraction (SVF) is administered to the patient suffering of Refractory Crohn's disease around of the fistula by local mico injection

SUMMARY:
Crohn's disease is a chronic inflammation of all or part of the digestive tract, " from the mouth to the anus ". .

Cell therapy is a new and promising approach for the treatment of inflammatory disease including Crohn's disease and fistulas.

Adipose tissue seems to be an ideal source for cell therapy. This is a prospective, open, non-comparative, single center, phase I-II clinical trial. It will involve 10 patients and will be conducted over a period of 28 month.

This protocol is designed to evaluate, in patients with Crohn's disease and fistula-in-ano refractory to conventional medical and surgical treatment, the safety and efficacy of local microinjection of autologous adipose tissue and SVF from microaspirate .

The main objective is to assess tolerance and security. The secondary objective is to evaluate the effectiveness of this technique

DETAILED DESCRIPTION:
Crohn's disease is a chronic inflammation of all or part of the digestive tract, " from the mouth to the anus ". Anoperineal lesions are a very frequent entity in this disease (20 to 80%) and a real therapeutic challenge. Among these lesions, we were interested in fistula-in-ano that are currently difficult to treat despite a large therapeutic arsenal.

Cell therapy is a new and promising approach for the treatment of inflammatory disease including Crohn's disease and fistulas.

Indeed, stem cells have shown some efficacy in several indications through their differentiation potential, including fistula-in-ano in Crohn's disease.

Adipose tissue seems to be an ideal source for cell therapy This is a prospective, open, non-comparative, single center, phase I-II clinical trial. It will involve 10 patients and will be conducted over a period of 28 month.

This protocol is designed to evaluate, in patients with Crohn's disease and fistula-in-ano refractory to conventional medical and surgical treatment, the safety and efficacy of local microinjection of autologous adipose tissue and SVF from microaspirate.

The main objective is to assess tolerance and security. The secondary objective is to evaluate the effectiveness of this technique Microaspiration is performed by a plastic surgeon under general anesthesia. He performs two types of fat removal : a sample of 120 cc wich is sent to the laboratory of cell therapy to obtain the SVF (5 cc) and a sample of 30 cc.

Once treatment obtained (SVF + adipose tissue) it is administered to the patient by local mico reinjection into (SVF) and around (adipose tissue) of the fistula. This administration is made by the surgeon under a second general anesthesia after viewing the fistula and removal of setons.

Then the patient is monitored with regular consultations at weeks 1, 2, 8, 16 et 48 and paraclinical (blood sample and magnetic resonance imaging of the perineum) at weeks 8 and 48 to evaluate tolerance and effectiveness of treatment.

At the end of the study, results that are expected are effectiveness of local micro reinjection of autologous adipose tissue and SVF for the treatment of refractory fistula-in-ano in Crohn's disease.

ELIGIBILITY:
Inclusion Criteria:

* Disease of Crohn diagnosed for at least 6 months according to the recognized clinical, endoscopic and histological criteria
* Presence of fistulas died anal complex estimated by clinical examination and MRI. A fistula died anal complex is, by definition, a fistula which answers at least one of the following criteria during its evolution: (1) high, trans-sphincter, extra-sphincter or above sphincter Inter-sphincter. (2) Presence of = 2 external openings. (3) Purulent Collections associated
* Active or slightly active Crohn luminal, defined by a CDAI (Crohn's Disease Activity Index) = 220

Exclusion Criteria:

- Disease of Crohn activates mainly luminal with a CDAI = 220 requiring an immediate treatment

* Patients having never received specific treatments of the anal died disease of Crohn with fistula, including by antibiotics
* Presence of an abscess or collections of more than 2 cms unless this problem is solved during the period of preparation
* Rectal and/or anal Stenosis and/or active proctitis, if it means a limitation of the surgical procedure
* Patient having undergone an operation of the fistula other than the drainage
* Patients under corticoids or by having receiving in the previous four weeks
* Active Malignant Tumors or history of Malignant tumors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-10; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
efficacy (measured as an absence of purulent collections superior to 2 cms concerning the fistula measured clinically and by MRI) | 48 weeks
  the patient is monitored with regular consultations at weeks 1, 2, 8, 16 et 48 and paraclinical (blood sample (hemogram , coagulation factors) and magnetic resonance imaging of the perineum) at weeks 8 and 48 to evaluate effectiveness of treatment. The efficacy of treatment is measured as an absence of purulent collections superior to 2 cms concerning the fistula treated at 12 and 48 weeks measured clinically and by MRI
safety (measured by an absence of fever and local inflammatories symptoms) | 48 weeks
  the patient is monitored with regular consultations at weeks 1, 2, 8, 16 et 48 and paraclinical (blood sample (hemogram and coagulation factors) and magnetic resonance imaging of the perineum) at weeks 8 and 48 to evaluate tolerance of treatment. The safety is measured by an absence of fever and local inflammatories symptoms measured at week 1, 2,8, 16 and 48

SECONDARY OUTCOMES:
improvement of quality of life (assessed by questionnaire) | 48 weeks
  Quality of life is assessed by questionnaire concerning (Inflammatory Bowel Disease) (SIBDQ: Short Inflammatory Bowel Disease Questionnaire) at week 2, 12, 16 et 48

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Charles GRIMAUD, MD, Principal Investigator — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France

REFERENCES:
- [Derived] Philandrianos C, Serrero M, Grimaud F, Magalon J, Visee C, Velier M, Francois P, Orsoni P, Magalon G, Grimaud JC, Desjeux A, Veran J, Sabatier F. First clinical case report of local microinjection of autologous fat and adipose-derived stromal vascular fraction for perianal fistula in Crohn's disease. Stem Cell Res Ther. 2018 Jan 10;9(1):4. doi: 10.1186/s13287-017-0736-6. PMID 29321063